CLINICAL TRIAL: NCT02157779
Title: Treatment of Trauma-Related Anger in OEF/OIF/OND Veterans
Acronym: TOTRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D1146-R; Rx 001146 (Other Grant/Funding Number: VA RR&D)
Record Dates: First submitted 2014-05-06; First posted 2014-06-06 (Estimated); Results first posted 2020-03-16 (Actual); Last update posted 2021-11-18 (Actual); Status verified 2021-10

CONDITIONS: Anger Problems
Keywords: Veterans; Anger; Cognitive Behavioral Therapy; Treatment

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cognitive Behavioral Intervention (CBI) (Experimental): 12 weekly individual sessions consisting of psychoeducation, and cognitive and behavioral anger management strategies
  Interventions: Behavioral: Cognitive Behavioral Intervention
- Supportive Intervention (SI) (Active Comparator): 12 weekly individual sessions consisting of psychoeducation, problem-solving strategies, and support
  Interventions: Behavioral: Supportive Intervention

INTERVENTIONS:
Behavioral: Cognitive Behavioral Intervention — Includes individual therapy sessions using cognitive and behavioral strategies addressing problems with anger intensity / frequency / management
  Other Names: CBI
  Arms: Cognitive Behavioral Intervention (CBI)
Behavioral: Supportive Intervention — Includes individual therapy sessions using supportive and problem-solving strategies.
  Arms: Supportive Intervention (SI)

SUMMARY:
Excessive and poorly controlled anger is one of the most common problems experienced by war Veterans. The consequences can be severe, including increased risk for divorce, domestic violence, job loss and instability, and other serious impairments in family, social, and occupational functioning. Availability of effective treatments is critical to reducing the adverse effects of anger in Veterans. The investigators propose to conduct a controlled study to determine whether a cognitive behavior treatment that has been adapted for treating anger problems in Veterans of Iraq and Afghanistan results in improved outcomes compared to a supportive therapy. Results will be examined for improvement in anger, functioning, and quality of life at end of 12 weekly sessions, and at 3 and 6 months following treatment.

DETAILED DESCRIPTION:
Poorly controlled anger is a common problem with often devastating effects in Veterans who have served in a warzone. Adverse consequences include increased risk for divorce, domestic violence, job loss and instability, and other serious impairments in family, social, and occupational functioning. Recent evidence indicates that anger and aggression are likely to be problems for a significant proportion of Veterans of Iraq (Operation Iraqi Freedom, OIF; Operation New Dawn, OND) and Afghanistan (Operation Enduring Freedom, OEF). A survey of reintegration problems among 754 OEF/OIF combat Veterans receiving VA Medical care showed that anger was the most commonly reported problem, with 57% reporting increased problems in controlling anger. Despite encouraging evidence for efficacy of cognitive behavioral interventions in treating anger in civilian samples, much less is known about the efficacy of such treatments for anger problems in military personnel following exposure to war zone trauma. Promising preliminary findings for individually based cognitive behavioral treatment have been reported, and there is evidence that a group anger management treatment delivered by teleconferencing is as effective as the same treatment delivered in person, but to date there is not a single adequately powered randomized trial designed to test the efficacy of an anger treatment compared to an active control condition in Veterans. Building on findings from the investigators' randomized pilot study, the objective of the current proposal is to conduct a randomized clinical trial with sufficient statistical power to test the effectiveness of a manualized cognitive behavioral intervention (CBI) that has been adapted from an existing treatment (Anger Control Therapy; Novaco, 1994, 2001) for the treatment of anger problems in OEF/OIF/OND Veterans, compared to a manualized supportive therapy intervention (SI) control condition. Ninety OEF/OIF/OND Veterans reporting significant problems with anger will be randomized to receive 12 individual sessions of one of the two study conditions. Outcomes including measures of anger and aggression; interpersonal, social and occupational functioning; and quality of life will be assessed during and at the end of treatment and at 3 and 6 month follow-ups. Exploratory analyses will examine 1) whether a diagnosis of PTSD impacts treatment effectiveness and 2) potential mediators of treatment outcome with CBI.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female current or former member of the military (active duty, National Guard or Reserve) Deployed to Iraq or Afghanistan
* Experience trauma during deployment
* Clinically significant anger
* At least 2 additional symptoms of PTSD hyperarousal
* If on medication, no changes within prior 4 weeks

Exclusion Criteria:

* Current severe substance use disorder or prior severe substance use disorder not in remission for at least 3 months
* Current psychotic symptoms
* current Mania or Bipolar Disorder
* Current suicidal or homicidal ideation requiring hospitalization
* Any severe cognitive impairment or history of Organic Mental Disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tracie M. Shea, PhD, Principal Investigator — Providence VA Medical Center, Providence, RI
Locations (1):
- Providence VA Medical Center, Providence, RI, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Yes
I anticipate sharing the data, but have not yet developed a specific plan.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: April 1 2021

REFERENCES:
- [Background] Shea MT, Lambert J, Reddy MK, Presseau C, Sevin E, Stout RL. Treatment of trauma related anger in operation enduring freedom, operation Iraqi freedom, and operation New Dawn veterans: Rationale and study protocol. Contemp Clin Trials Commun. 2018 Aug 24;12:26-31. doi: 10.1016/j.conctc.2018.08.011. eCollection 2018 Dec. PMID 30225391

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from a wide range of sources during the time period of January 1, 2015 through January 31, 2018. The primary recruitment source was the Providence Veterans Affairs Medical Center, including the OEF/OIF specialty primary care clinic, the Returning Veterans Outreach Program (REVOC) and the PTSD Clinic.
Pre-assignment Details: Of the 112 enrolled, 94 completed both the first and second baseline assessments and were deemed eligible for the study. Of the 94 who completed their second baseline and were deemed eligible for the study, 92 were randomized to treatment. Two of the 92 randomized participants did not respond to outreach and did not start treatment.
Groups:
- Cognitive Behavioral Intervention: 12 weekly individual sessions consisting of psychoeducation, and cognitive and behavioral anger management strategies
  Cognitive Behavioral Intervention: Includes individual therapy sessions using cognitive and behavioral strategies addressing problems with anger intensity / frequency / management
- Supportive Intervention: 12 weekly individual sessions consisting of psychoeducation, problem-solving strategies, and support
  Supportive Intervention: Includes individual therapy sessions using supportive and problem-solving strategies.
Period: Overall Study
Arm/Group | Cognitive Behavioral Intervention | Supportive Intervention
Started | 47 | 45
Completed | 23 | 34
Not Completed | 24 | 11
Not completed — Logistical | 9 | 3
Not completed — Stopped attending, reason unknown | 11 | 7
Not completed — No response to outreach after Baseline | 1 | 1
Not completed — Moved | 1 | 0
Not completed — Medical | 1 | 0
Not completed — Legal issue | 1 | 0

BASELINE CHARACTERISTICS:
Population: Number of participants varies slightly for some measures due to missing data.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cognitive Behavioral Intervention | Supportive Intervention | Total
Number analyzed (Participants) | 47 | 45 | 92
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.30 (9.11) | 36.5 (9.77) | 35.90 (9.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 46 | 43 | 89
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 12 | 19
  Not Hispanic or Latino | 40 | 33 | 73
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 3 | 4
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 4 | 5
  White | 42 | 35 | 77
  More than one race | 2 | 3 | 5
  Unknown or Not Reported | 0 | 0 | 0
Employment Status [Count of Participants; unit: Participants]
  Full Time | 22 | 27 | 49
  Part Time | 5 | 15 | 20
  Unemployed | 14 | 3 | 17
  Retired | 6 | 0 | 6
Education [Count of Participants; unit: Participants]
  High School Graduate/GED | 11 | 11 | 22
  Some College/Technical School | 30 | 24 | 54
  College Graduate | 4 | 7 | 11
  Post Graduate | 2 | 3 | 5
State Trait Anger Inventory 2 (STAXI-2) Anger Expression Index Score [Mean (Standard Deviation); unit: units on a scale] — STAXI-2 is a self-report questionnaire consisting of six scales and an Anger Expression Index. The Anger Expression Index is an overall measure of the expression and control of anger based on responses to two anger expression and two anger control subscales. Score range is 0 to 96; higher scores means more anger.
  units on a scale | 55.67 (12.98) | 54.77 (11.86) | 55.24 (12.39)
Overt Anger Scale-Modified Aggression Scale [Mean (Standard Deviation); unit: units on a scale] — Structured Interview that assesses verbal and physical aggressive behaviors. Four subscores are calculated by multiplying frequency by severity of specific behaviors within that category. Subscores are also weighted for severity. The Aggression Scale Score is the total of subscores. Minimum score is zero; no maximum score specified as scores are determined by unlimited frequency counts of behavior. Higher scores indicate more frequent and severe aggressive behaviors.
  units on a scale | 1.335 (0.525) | 1.396 (0.500) | 1.365 (0.511)
Longitudinal Interval Follow up (LIFE) social functioning global score [Mean (Standard Deviation); unit: units on a scale] — LIFE psychosocial functioning scales assess functioning in multiple areas, including work, interpersonal relationships, recreation, and global social adjustment. The global social adjustment score ranges from 1 to 5, with higher scores reflecting poorer functioning.
  units on a scale | 3.57 (0.54) | 3.64 (0.71) | 3.61 (0.63)
LIFE Work Functioning Global Score [Mean (Standard Deviation); unit: units on a scale] — The LIFE Work Functioning Score assess functioning in work (employment, household, or student). The work global score ranges from 1 to 5; higher scores indicate worse functioning.
  units on a scale | 3.17 (1.22) | 2.98 (1.08) | 3.08 (1.15)
Outcomes Questionnaire [Mean (Standard Deviation); unit: units on a scale] — The Outcomes questionnaire is a self report measure that assesses functioning and includes three subscales: symptom distress, interpersonal relations, and social role functioning. The total score is the sum of the scores for the three scales. Total scores can range from 0 to 180; higher scores mean worse functioning.
  units on a scale | 82.45 (26.50) | 88.31 (22.93) | 85.32 (24.86)
WHO Quality of Life (WHOQOL) Psychological Domain [Mean (Standard Deviation); unit: units on a scale] — The WHOQOL is a 26 item self report measure used to assess quality of life in multiple domains. The psychological domain includes 6 items, each rated on a scale from 1 to 5. The score is obtained by computing the means of each item of the scale, and multiplying the mean by 4. Scores can range from 4 to 20. Higher scores reflect better quality of life.
  units on a scale | 11.54 (3.17) | 10.97 (2.61) | 11.26 (2.91)
Clinician Administered PTSD Scale (CAPS) [Mean (Standard Deviation); unit: units on a scale] — The CAPS-5 is a clinician administered structured interview assessing the DSM-5 PTSD symptoms. Each of the 20 symptoms is rated on a 0 to 4 scale; the range for the total score is 0 to 80. Higher scores reflect more severe PTSD.
  units on a scale | 30.02 (10.62) | 32.38 (9.52) | 31.17 (10.11)

OUTCOME MEASURES:

1. Primary Outcome: Least Squares Mean Anger Expression Index Score on the State Trait Anger Inventory 2 (STAXI-2) Using a Repeated Measures ANCOVA Adjusted for Baseline and Time Effects
Description: The STAXI-2 is a revision of Spielberger's State-Trait Anger Expression Inventory (STAXI), expanded from 44 to 57 items. It is a self-report questionnaire consisting of six scales and an Anger Expression Index (AX). Scales include State Anger, Trait Anger, Anger Expression-Out, Anger Expression-In, Anger Control-Out and Anger Expression-In. The Anger Expression Index is an overall measure of the expression and control of anger based on responses to the two anger expression and the two anger control subscales. Minimum and Maximum Values range from 0 to 96, higher scores mean more anger.
Time Frame: Baseline, Weeks 4, 8,12, 3 and 6 months post-treatment
Population: Participants were randomly assigned to CBI or SI. Those with one or more post-baseline assessments were included in Hierarchical Linear Model (HLM) analyses. Not all participants had post-baseline data; some treatment noncompleters had one or more post-baseline assessments. Least Square Means and differences adjusted for baseline and time effects from repeated measures ANCOVA are shown. Full Information Maximum Likelihood was used to account for missing data.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Cognitive Behavioral Intervention (CBI) | Supportive Intervention (SI)
Number analyzed (Participants) | 32 | 35
score on a scale | 41.42 (1.77) | 47.09 (1.65)
Statistical Analysis 1: Comparison: Cognitive Behavioral Intervention (CBI) vs Supportive Intervention (SI); All randomized participants with at least one post-baseline assessment (4wk, 8wk, end of treatment, 3 mo f/u, and/or 6 mo f/u) were used in the HLM analyses; Test type: Superiority; p = .017, ANCOVA — Threshold for statistical significance was 0.025; Method used: Hierarchical Linear Model (HLM) Repeated Measures Analysis of Covariance, Controlling for Baseline Score; Least Squares Mean Difference = -5.68, 95% CI 2-sided [-10.32 to -1.01] — A negative difference means that the adjusted mean for CBI is numerically lower than that for SI

2. Primary Outcome: Least Squares Mean Aggression Scale Score on the Overt Aggression Scale-Modified (OAS-M) Using a Repeated Measures ANCOVA Adjusted for Baseline Scores and Time Effects
Description: Structured Interview that assesses verbal and physical aggressive behaviors. Minimum and Maximum Values range from 0 to no maximum, higher scores mean more anger.
Time Frame: Baseline, Weeks 4, 8,12 (end of treatment), 3 and 6 months post-treatment
Population: Participants were randomly assigned to CBI or SI. Participants with at least one post-baseline measure (4wk, 8wk, 12 wk, 3 mo and/or 6 mo f/u) were included in HLM analysis. Not all participants had post-baseline data, and some non-completers had one or more post-baseline assessments. Least Square means and differences adjusted for baseline and time effects from repeated analyses of covariance are shown. Full Information Maximum Likelihood was used to account for missing data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Cognitive Behavioral Intervention | Supportive Intervention
Number analyzed (Participants) | 34 | 39
units on a scale | 1.00 (0.08) | 1.14 (0.07)
Statistical Analysis 1: Comparison: Cognitive Behavioral Intervention vs Supportive Intervention; Population Description: All randomized participants with at least one post-baseline assessment (4wk, 8wk, end of treatment, 3 mo f/u, and/or 6 mo f/u) were used in the statistical analysis. Data were winsorized and log10 transformed to counter high levels of skewness. Full Information Maximum Likelihood was used to account for missing data; Test type: Superiority; p = 0.19, ANCOVA — The threshold for statistical significance was p=0.025; Hierarchical Linear Model (HLM) Repeated Measures Analysis of Covariance, Controlling for Baseline Score; Least Squares Mean Difference = -0.14, 95% CI 2-sided [-0.33 to 0.06]; A negative difference means that the adjusted mean for CBI is numerically lower than that for SI

3. Secondary Outcome: Least Squares Mean Global Social Adjustment Score on the Longitudinal Interval Follow-up Evaluation (LIFE) Using a Repeated Measures ANCOVA Adjusted for Baseline Scores and Time Effects
Description: Psychosocial functioning scales from the clinician administered Longitudinal Interval Follow-up Evaluation (LIFE) provides assessment of functioning in areas of work (employment, household, or student), various aspects of interpersonal functioning, recreation and satisfaction. The global social adjustment score is based upon a 5 point scale. Ratings are based on the past month. The psychosocial functioning ratings have been found to be of generally high reliability. Minimum and Maximum Values range from 1 to 5, higher scores mean worse functioning.
Time Frame: Baseline, 12 weeks (end of treatment), 3 and 6 months post-treatment
Population: Participants were randomly assigned to CBI or SI. Those with at least one post-baseline measure (12 wk (end of treatment), 3 mo f/u, and/or 6 mo f/u) were included in HLM analysis. Not all had post-baseline data, and some who didn't complete treatment had one or more post-baseline assessments. Least Square means and differences adjusted for baseline and time effects from repeated measures ANCOVA are shown. Full Information Maximum Likelihood was used to account for missing data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Cognitive Behavioral Intervention | Supportive Intervention
Number analyzed (Participants) | 27 | 37
units on a scale | 2.85 (0.13) | 3.28 (0.10)
Statistical Analysis 1: Comparison: Cognitive Behavioral Intervention vs Supportive Intervention; Population Description: All randomized participants with at least one post-baseline assessment were used in the statistical analysis process; Test type: Superiority; p = .011, ANCOVA — Threshold for statistical significance was 0.025; Hierarchical Linear Model (HLM) Repeated Measures Analysis of Covariance, Controlling for Baseline Score; Least Squares Mean Difference = -0.42, 95% CI 2-sided [-0.75 to -0.09]; A negative difference means that the adjusted mean for CBI is numerically lower than that for SI

4. Secondary Outcome: Least Squares Mean Global Work Functioning Score on the Longitudinal Interval Follow-up Evaluation (LIFE) Using a Repeated Measures ANCOVA Adjusted for Baseline Scores and Time Effects
Description: Psychosocial functioning scales from the clinician administered Longitudinal Interval Follow-up Evaluation (LIFE) provides assessment of functioning in areas of work (employment, household, or student), various aspects of interpersonal functioning, recreation, satisfaction and global social adjustment. Ratings are based on the past month. The psychosocial functioning ratings have been found to be of generally high reliability. Minimum and Maximum Values for the work functioning global score range from 1 to 5, higher scores mean worse functioning.
Time Frame: Baseline, 12 weeks (end of treatment), 3 and 6 months post-treatment
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Cognitive Behavioral Intervention | Supportive Intervention
Number analyzed (Participants) | 27 | 37
units on a scale | 2.78 (0.14) | 3.04 (0.12)
Statistical Analysis 1: Comparison: Cognitive Behavioral Intervention vs Supportive Intervention; All randomized participants with at least one post-baseline assessment (12 weeks (end of treatment, 3 month and/or 6 month follow-up) were included in the analyses; Test type: Superiority; p = 0.16, ANCOVA — Threshold for statistical significance was 0.025; Hierarchical Linear Model (HLM) Repeated Measures Analysis of Covariance, Controlling for Baseline Score; Least Squares Mean Difference = -0.26, 95% CI 2-sided [-0.63 to 0.11] — A negative difference means that the adjusted mean for CBI is numerically lower than that for SI

5. Secondary Outcome: Least Squares Mean Total Score on the Outcomes Questionnaire (OQ) Using a Repeated Measures ANCOVA Adjusted for Baseline Scores and Time Effects
Description: The OQ is a self report measure that assesses functioning and includes three subscales: symptom distress, interpersonal relations, and social role functioning. Concurrent validity has been demonstrated in relation to internal consistency and reliability. Additionally, the OQ has been shown to be fairly stable in untreated individuals and sensitive to change in those individuals in treatment. Minimum and Maximum Values range from 0 to 180, higher scores mean worse functioning.
Time Frame: Baseline, 12 weeks, 3 and 6 months post-treatment
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Cognitive Behavioral Intervention | Supportive Intervention
Number analyzed (Participants) | 26 | 37
score on a scale | 60.69 (4.11) | 72.34 (3.27)
Statistical Analysis 1: Comparison: Cognitive Behavioral Intervention vs Supportive Intervention; All randomized participants with at least one post-baseline assessment (12 weeks (end of treatment), 3 month and/or 6 month follow-up) were included in the statistical analyses; Test type: Superiority; p = .031, ANCOVA — Threshold for statistical significance was 0.025; Hierarchical Linear Model (HLM) Repeated Measures Analysis of Covariance, Controlling for Baseline Score; Least Squares Mean Difference = -11.65, 95% CI 2-sided [-22.20 to -1.09] — A negative difference means that the adjusted mean for CBI is numerically lower than that for SI

6. Secondary Outcome: Least Squares Mean Psychological Domain Score on the WHO Quality of Life (WHOQOL) Using a Repeated Measures ANCOVA Adjusted for Baseline Scores and Time Effects
Description: The World Health Organization Quality of Life (WHOQOL-BREF), is 26 item self-report measure used to assess quality of life in multiple domains (i.e., physical, psychological, social, and environment). Psychometric properties suggest that the measure is valid and reliable across cultures and nations. Ratings are made on a 5 point scale. The psychological subscale, which consists of 6 items, was used in this study. Minimum and Maximum Values for the psychological domain range from 6 to 30, higher scores mean better quality of life.
Time Frame: Baseline, 12 weeks (end of treatment), 3 and 6 months post-treatment
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Cognitive Behavioral Intervention | Supportive Intervention
Number analyzed (Participants) | 25 | 35
score on a scale | 13.64 (0.40) | 12.09 (0.33)
Statistical Analysis 1: Comparison: Cognitive Behavioral Intervention vs Supportive Intervention; All randomized participants with at least one post-baseline assessment (week 12 (end of treatment), 3 month, and/or 6 month follow-up) were used in the statistical analysis; Test type: Superiority; p = 0.004, ANCOVA — Threshold for statistical significance was 0.025; Hierarchical Linear Model (HLM) Repeated Measures Analysis of Covariance, Controlling for Baseline Score; Least Squares Mean Difference = 1.56, 95% CI 2-sided [0.51 to 2.60]; A positive difference means that the adjusted mean for CBI is numerically higher than that for SI

7. Secondary Outcome: Least Squares Mean PTSD Severity Score on the Clinician-Administered PTSD Scale (CAPS) for DSM-5 Using a Repeated Measures ANCOVA Adjusted for Baseline Scores and Time Effects
Description: The CAPS-5 (updated for DSM-5) is a clinician administered structured interview for the assessment of DSM-5 PTSD. The CAPS has excellent reliability and validity and is widely used in PTSD treatment research. Each one of the DSM-5 PTSD symptoms is rated on a 0-4 (low to high) scale to determine symptom severity. The cutoff used to establish the presence of an individual symptom is a score of 2 or greater. Overall PTSD severity is computed by summing the totals for all items. Minimum and Maximum Values range from 0 to 80, higher scores mean higher levels of symptomatology.
Time Frame: Baseline,12 weeks (end of treatment), 3 and 6 months post-treatment
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Cognitive Behavioral Intervention | Supportive Intervention
Number analyzed (Participants) | 27 | 37
score on a scale | 22.56 (2.01) | 24.71 (1.69)
Statistical Analysis 1: Comparison: Cognitive Behavioral Intervention vs Supportive Intervention; All randomized participants with at least one post-baseline assessment were used in the statistical analysis process; Test type: Superiority; p = 0.416, ANCOVA — Threshold for statistical significance was 0.025; Hierarchical Linear Model (HLM) Repeated Measures Analysis of Covariance, Controlling for Baseline Score; Least Squares Mean Difference = -2.15, 95% CI 2-sided [-7.37 to 3.07] — A negative difference means that the adjusted mean for CBI is numerically lower than that for SI

8. Other Pre Specified Outcome: Least Squares Mean Total Score on the Anger Consequences Questionnaire (ACQ) Using a Repeated Measures ANCOVA Adjusted for Baseline Scores and Time Effects
Description: The ACQ is a brief self-report measure developed to assess the frequency of negative anger-related behavioral consequences. Internal consistencies of .75 to .91 have been reported. This scale includes items not covered by the other anger measures, including for example, trouble with the law, driving recklessly, getting into an accident, damaging relationships, etc. There are 50 items; minimum and maximum Values range from 0 to 200. Higher scores means more anger.
Time Frame: Baseline, Week 12, 3 and 6 months Post-treatment
Population: Participants were randomly assigned to CBI or SI. Those with one or more post-baseline assessments (week 12, 3- and/or 6-month follow-up) were included in HLM analyses. Not all participants had post-baseline data, and some who didn't complete treatment had one or more post-baseline assessments. Least Square means and differences adjusted for baseline and time effects from repeated measures ANCOVA are shown. Full Information Maximum Likelihood was used to account for missing data.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Cognitive Behavioral Intervention (CBI) | Supportive Intervention (SI)
Number analyzed (Participants) | 25 | 35
score on a scale | 30.48 (4.71) | 44.20 (3.75)
Statistical Analysis 1: Comparison: Cognitive Behavioral Intervention (CBI) vs Supportive Intervention (SI); All randomized participants with at least one post-baseline assessment were used in the analyses; Test type: Superiority; p = 0.028, ANCOVA — Threshold for significance was 0.025; Hierarchical Linear Model (HLM) Repeated Measures Analysis of Covariance controlling for baseline score; Least Squares Mean Difference = -13.72, 95% CI 2-sided [-25.94 to -1.50] — A negative difference means that the adjusted mean for CBI is numerically lower than that for SI

9. Post Hoc Outcome: Mean Scores for Sessions 1-4, 5-8, and 9-12 on the Dimensions of Anger Response (DAR) Measure Using a Generalized Linear Model (GLM) Repeated Measures ANOVA
Description: The DAR is a 7 item self-report measure of anger reactions. It has been found to be reliable and sensitive to change. Higher scores reflect more severe anger. Scores can range from 0 to 28.
Time Frame: The DAR was administered at each weekly 75-minute treatment session (up to 12 sessions). The mean DAR scores for sessions 1-4, 5-8, and 9-12 were calculated and used as outcome variables in the GLM repeated measures ANOVA.
Population: Participants were randomly assigned to CBI or SI. Participants with at one or more DARs completed during each of the time frames (sessions 1-4, 5-8, 9-12) were included in the analyses. Not all randomized participants had one or more DARs in all time frames. Some who did not complete treatment did have at least one DAR in all time frames.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Behavioral Intervention | Supportive Intervention
Number analyzed (Participants) | 25 | 34
score on a scale
  Sessions 1-4 | 14.35 (4.91) | 15.43 (5.65)
  Sessions 5-8 | 10.76 (5.77) | 12.96 (5.99)
  Sessions 9-12 | 8.60 (5.80) | 11.88 (6.53)
Statistical Analysis 1: Comparison: Cognitive Behavioral Intervention vs Supportive Intervention; All randomized participants with at least one DAR completed in each time frame (sessions 1-4, 5-8, and 9-12) were included in the analyses. The mean DAR scores for sessions 1-4, 5-8, and 9-12 were calculated and used as outcome variables in the GLM repeated measures ANOVA; Test type: Superiority; p = 0.13, ANOVA; GLM Repeated Measures Analysis of Variance of means grouped by sessions 1-4, 5-8, and 9-12

10. Post Hoc Outcome: Least Squares Mean Global Anger and Aggression Score on the Overt Aggression Scale-Modified (OAS-M) Using a Repeated Measures ANCOVA Adjusted for Baseline Scores and Time Effects
Description: The OAS-M is a structured Interview that assesses verbal and physical aggressive behaviors. The Global Anger and Aggression Score consists of two items - subjective experience and overt expression of anger, each rated on a scale from 0 to 5. Minimum and Maximum Values range from 0 to 10, higher scores means more anger.
Time Frame: Baseline, Weeks 4, 8,12, 3 and 6 months post-treatment
Population: Participants were randomly assigned to the CBI or SI. Those with at least one post-baseline measure (4wk, 8wk, 12 wk, 3 mo and/or 6 mo f/u) were included in HLM analysis. . Not all participants had post-baseline data, and some non-completers had one or more post-baseline assessments. Least Square means and differences adjusted for baseline and time effects from repeated analyses of covariance are shown. Full Information Maximum Likelihood was used to account for missing data.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Cognitive Behavioral Intervention | Supportive Intervention
Number analyzed (Participants) | 34 | 39
score on a scale | 4.02 (0.29) | 4.84 (0.26)
Statistical Analysis 1: Comparison: Cognitive Behavioral Intervention vs Supportive Intervention; All randomized participants with at least one post-baseline assessment (week 4, week 8, week 12 (end of treatment), 3 mo and/or 6 month follow-up) were included in the HLM analyses; Test type: Superiority; p = 0.030, ANCOVA — Threshold for statistical significance was 0.025; Hierarchical Linear Model (HLM) Repeated Measures Analysis of Covariance, Controlling for Baseline Score; Least Squares Mean Difference = -0.82, 95% CI 2-sided [-1.578 to -0.063] — A negative difference means that the adjusted mean for CBI is numerically lower than that for SI

11. Post Hoc Outcome: Least Squares Mean Aggressive Outbursts Score From the Overt Aggression Scale-Modified (OAS-M) Using a Repeated Measures ANCOVA Adjusted for Baseline Scores and Time Effects
Description: The OAS-M is a structured Interview that assesses verbal and physical aggressive behaviors. Aggressive Outbursts is a measure of the frequency and severity of all aggressive outbursts over the past week.Minimum and Maximum Values range from 0 to no maximum, higher scores means more anger.
Time Frame: Baseline, Weeks 4, 8,12, 3 and 6 months post-treatment
Population: Participants were randomly assigned to CBI or SI. Participants with at least one post-baseline measure (4wk, 8wk, 12 wk, 3 mo and/or 6 mo f/u) were included in HLM analysis. Not all had post-baseline data, and some who didn't complete treatment had one or more post-baseline assessments. Least Square means and differences adjusted for baseline and time effects from repeated measures ANCOVA are shown. Full Information Maximum Likelihood was used to account for missing data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Cognitive Behavioral Intervention | Supportive Intervention
Number analyzed (Participants) | 34 | 39
units on a scale | 0.26 (0.03) | 0.34 (0.02)
Statistical Analysis 1: Comparison: Cognitive Behavioral Intervention vs Supportive Intervention; All randomized participants with at least one post-baseline assessment (4 week, 8 week, 12 week, 3 month and/or 6 month follow-up) were included in the HLM analysis. Data were winsorized and log10 transformed to counter high levels of skewness. Full Information Maximum Likelihood was used to account for missing data; Test type: Superiority; p = 0.021, ANCOVA — Threshold for statistical significance was 0.025; Hierarchical Linear Model (HLM) Repeated Measures Analysis of Covariance, Controlling for Baseline Score; Least Squares Mean Difference = -0.085, 95% CI 2-sided [-0.158 to -0.011] — A negative difference means that the adjusted mean for CBI is numerically lower than that for SI

12. Post Hoc Outcome: Least Squares Mean Verbal Assault Score on the Overt Aggression Scale-Modified (OAS-M) Using a Repeated Measures ANCOVA Adjusted for Baseline Scores and Time Effects
Description: The OAS-M is a structured interview that assesses frequency of anger and aggression. The verbal assault subscale measures the frequency and severity of verbal assaults over the previous week. Minimum and Maximum Values range from 0 to no maximum, higher scores means more anger.
Time Frame: Baseline, 4 weeks, 8 weeks, 12 weeks (end of treatment), 3 month and 6 month follow-ups
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Cognitive Behavioral Intervention | Supportive Intervention
Number analyzed (Participants) | 34 | 39
units on a scale | 0.85 (0.07) | 0.96 (0.06)
Statistical Analysis 1: Comparison: Cognitive Behavioral Intervention vs Supportive Intervention; All randomized participants with at least one post-baseline assessment (4 week, 8 week, 12 week, 3 month and/or 6 month follow-up) were used in the HLM analysis. Data were winsorized and log10 transformed to counter high levels of skewness. Full Information Maximum Likelihood was used to account for missing data; Test type: Superiority; p = 0.246, ANCOVA — Threshold for significance was 0.025; Hierarchical Linear Model (HLM) Repeated Measures Analysis of Covariance, Controlling for Baseline Score; Least Squares Mean Difference = -0.10, 95% CI 2-sided [-0.283 to 0.073] — A negative difference means that the adjusted mean for CBI is numerically lower than that for SI

13. Post Hoc Outcome: Least Squares Mean Assaults on Objects Score on the Overt Aggression Scale-Modified (OAS-M) Using a Repeated Measures ANCOVA Adjusted for Baseline Scores and Time Effects
Description: The OAS-M is a structured interview that assesses anger and aggressive behaviors. The Assaults on Objects Subscale assesses the frequency and severity of assaults against objects over the past week. Minimum and Maximum Values range from 0 to no maximum, higher scores means more assaults.
Time Frame: Baseline, weeks 4, 8, 12 (post-treatment), 3 and 6 month post-treatment follow-ups
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Cognitive Behavioral Intervention | Supportive Intervention
Number analyzed (Participants) | 34 | 39
units on a scale | 0.19 (0.05) | 0.33 (0.04)
Statistical Analysis 1: Comparison: Cognitive Behavioral Intervention vs Supportive Intervention; All randomized participants with at least one post-baseline assessment were used in the statistical analysis. Data were winsorized and log 10 transformed to counter high levels of skewness; Test type: Superiority; p = 0.036, ANCOVA — Threshold for statistical significance was 0.025; Hierarchical Linear Model (HLM) Repeated Measures Analysis of Covariance, Controlling for Baseline Score; Least Squares Mean Difference = -0.14, 95% CI 2-sided [-0.27 to -0.01] — A negative difference means that the adjusted mean for CBI is numerically lower than that for SI

14. Post Hoc Outcome: Least Squares Mean Assault Against Others Score on the Overt Aggression Scale-Modified Using a Repeated Measures ANCOVA Adjusted for Baseline Scores and Time Effects
Description: The Assault Against Others Subscale assesses the frequency and severity of aggressive behaviors towards others. Minimum and Maximum Values range from 0 to no maximum, higher scores means more anger.
Time Frame: Baseline, weeks 4, 8, 12 (post-treatment), 3 and 6 month post-treatment
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Cognitive Behavioral Intervention | Supportive Intervention
Number analyzed (Participants) | 34 | 39
units on a scale | 0.11 (0.06) | 0.14 (0.05)
Statistical Analysis 1: Comparison: Cognitive Behavioral Intervention vs Supportive Intervention; [analysis description as in outcome 11, analysis 1]; Test type: Superiority; p = 0.786, ANCOVA — Threshold for statistical significance was 0.025; Hierarchical Linear Model (HLM) Repeated Measures Analysis of Covariance, controlling for baseline score; Least Squares Mean Difference = -0.026, 95% CI 2-sided [-0.213 to 0.1614] — A negative difference means that the adjusted mean for CBI is numerically lower than that for SI

15. Post Hoc Outcome: Least Squares Mean Assault Against Self Scale on the Overt Aggression Scale-Modified Using a Repeated Measures ANCOVA Adjusted for Baseline Scores and Time Effects
Description: The OAS-M is a structured interview assessing anger and aggression. The Assault against Self Subscale assesses the frequency and severity of aggression towards oneself during the past week. Minimum and Maximum Values range from 0 to no maximum, higher scores means more anger.
Time Frame: Baseline, weeks 4, 8, 12 (posttreatment), 3 and 6 months posttreatment
Population: All randomized participants with at least one post-baseline assessment (4wk, 8wk, end of treatment, 3 mo f/u, and/or 6 mo f/u) were included in the analyses. Data were winsorized and log 10 transformed to counter high levels of skewness. Least Square means and differences adjusted for baseline and time effects from repeated analyses of covariance are shown. Full Information Maximum Likelihood was used to account for missing data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Cognitive Behavioral Intervention | Supportive Intervention
Number analyzed (Participants) | 34 | 39
units on a scale | 0.11 (0.06) | 0.14 (0.05)
Statistical Analysis 1: Comparison: Cognitive Behavioral Intervention vs Supportive Intervention; [analysis description as in outcome 11, analysis 1]; Test type: Superiority; p = 0.744, ANCOVA — Threshold for significance was 0.025; Hierarchical Linear Model (HLM) Repeated Measures Analysis of Covariance, controlling for baseline score; Least Squares Mean Difference = -0.02, 95% CI 2-sided [-0.18 to 0.13] — A negative difference means that the adjusted mean for CBI is numerically lower than that for SI

16. Post Hoc Outcome: Least Squares Mean Anger Expression Out Scale Score on the State Trait Anger Inventory 2 (STAXI-2) Using a Repeated Measures ANCOVA Adjusted for Baseline Scores and Time Effects
Description: The revised STAXI-2 is a 57 item self-report questionnaire that consists of five subscales and an anger expression index. The Anger Expression Out (AX-O) subscale measures how often angry feelings are expressed in verbally or physically aggressive behavior. It consists of 8 items, with a subscale range of 8 to 32. Higher scores indicate higher levels of expressed anger.
Time Frame: Baseline, weeks 4, 8, 12 (post-treatment), 3 and 6 month post-treatment
Population: Participants were randomly assigned to CBI or SI. Those with at least one post-baseline measure (4 wk, 8wk,12 wk (end of tx), 3 mo and/or 6 mo f/u) were included in HLM analysis. Not all had post-baseline data, and some who didn't complete treatment had one or more post-baseline assessments. Least Square means and differences adjusted for baseline and time effects from repeated measures ANCOVA are shown. Full Information Maximum Likelihood was used to account for missing data.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Cognitive Behavioral Intervention | Supportive Intervention
Number analyzed (Participants) | 33 | 36
score on a scale | 16.42 (0.44) | 18.27 (0.41)
Statistical Analysis 1: Comparison: Cognitive Behavioral Intervention vs Supportive Intervention; All randomized participants with at least one post-baseline assessment (4 week, 8 week, 12 week, 3 month and/or 6 month follow-up) were included in the HLM analysis. Full Information Maximum Likelihood was used to account for missing data; Test type: Superiority; p = 0.002, ANCOVA — Threshold for significance was 0.025; Hierarchical Linear Model (HLM) Repeated Measures Analysis of Covariance, controlling for baseline score; Least Squares Mean Difference = -1.85, 95% CI 2-sided [-3.038 to -0.663] — A negative difference means that the adjusted mean for CBI is numerically lower than that for SI

17. Post Hoc Outcome: Least Squares Mean Anger Expression Scale Score on the State-Trait Anger Inventory Using a Repeated Measures ANCOVA Adjusted for Baseline Scores and Time Effects
Description: The revised STAXI-2 is a 57 item self-report questionnaire that consists of five subscales and an anger expression index. The Anger Expression In subscale measures how often angry feelings are experienced but not expressed (suppressed). It consists of 8 items with a score range of 8-32. Higher scores indicate higher levels of experienced anger.
Time Frame: Baseline, weeks 4, 8, 12 (post-treatment), 3 and 6 month post-treatment
Population: Participants were randomly assigned to CBI or SI. Those with at least one post-baseline measure (4 wk, 8 wk, 12 wk (posttreatment), 3 mo and/or 6 mo f/u) were included in HLM analysis. Not all had post-baseline data, and some who didn't complete treatment had one or more post-baseline measures. Least Square means and differences adjusted for baseline and time effects from repeated measures ANCOVA are shown. Full Information Maximum Likelihood was used to account for missing data.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Cognitive Behavioral Intervention | Supportive Intervention
Number analyzed (Participants) | 33 | 36
score on a scale | 18.31 (0.55) | 19.31 (0.52)
Statistical Analysis 1: Comparison: Cognitive Behavioral Intervention vs Supportive Intervention; All randomized participants with at least one post-baseline assessment (4wk, 8wk, 12 week (end of treatment), 3 mo and/or 6 mo follow-up) were included in the HLM analysis. Full Information Maximum Likelihood was used to account for missing data; Test type: Superiority; p = 0.186, ANCOVA — Threshold for significance was 0.025; Hierarchical Linear Model (HLM) Repeated Measures Analysis of Covariance, controlling for baseline score; Least Squares Mean Difference = -1.0, 95% CI 2-sided [-2.518 to 0.524] — A negative difference means that the adjusted mean for CBI is numerically lower than that for SI

18. Post Hoc Outcome: Least Squares Mean Score on the Anger Control Out Scale From the State Trait Anger Inventory-2 (STAXI-2) Using a Repeated Measures ANCOVA Adjusted for Baseline Scores and Time Effects
Description: The STAXI-2 Anger Control Out subscale measures how often a person controls the outward expression of angry feelings. It consists of 8 items with a score range of 8 to 32. Higher scores reflect more effort in monitoring and preventing the outward expression of anger.
Time Frame: Baseline, weeks 4, 8, 12 (post-treatment), 3 and 6 month post-treatment Baseline, weeks 4, 8, 12 (post-treatment), 3 and 6 month post-treatment
Population: Participants were randomly assigned to CBI or SI. Those with at least one post-baseline measure (posttreatment), 3 mo and/or 6 mo f/u) were included in HLM analysis. Not all had post-baseline data, and some who didn't complete treatment had one or more post-baseline measures. Least Square means and differences adjusted for baseline and time effects from repeated measures ANCOVA are shown. Full Information Maximum Likelihood was used to account for missing data.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Cognitive Behavioral Intervention | Supportive Intervention
Number analyzed (Participants) | 32 | 36
score on a scale | 20.07 (0.68) | 18.80 (0.62)
Statistical Analysis 1: Comparison: Cognitive Behavioral Intervention vs Supportive Intervention; [analysis description as in outcome 17, analysis 1]; Test type: Superiority; p = 0.164, ANCOVA — Threshold for significance was 0.025; Hierarchical Linear Model (HLM) Repeated Measures Analysis of Covariance, controlling for baseline score; Least Squares Mean Difference = 1.26, 95% CI 2-sided [-0.560 to 3.09] — A positive difference means that the adjusted mean for CBI is numerically higher than that for SI

19. Post Hoc Outcome: Least Squares Mean Anger Control-In Score on the State-Trait Anger Expression Inventory-2 (STAXI-2) Using a Repeated Measures ANCOVA Adjusted for Baseline Scores and Time Effects
Description: The STAXI-2 Anger Control-In subscale measures how often a person attempts to control angry feelings by calming down or cooling off. It has 8 items with a score range of 8 to 32. Higher scores indicate more frequent attempts to control internal experiences of anger.
Time Frame: Baseline, weeks 4, 8, 12 (post-treatment), 3 and 6 month post-treatment
Population: as for outcome 17
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Cognitive Behavioral Intervention | Supportive Intervention
Number analyzed (Participants) | 33 | 36
score on a scale | 20.71 (0.68) | 19.38 (0.54)
Statistical Analysis 1: Comparison: Cognitive Behavioral Intervention vs Supportive Intervention; [analysis description as in outcome 17, analysis 1]; Test type: Superiority; p = 0.100, ANCOVA — Threshold for statistical significance was 0.025; Hierarchical Linear Model (HLM) Repeated Measures Analysis of Covariance, Controlling for Baseline Score; Least Squares Mean Difference = 1.33, 95% CI 2-sided [-0.26 to 2.92] — A positive difference means that the adjusted mean for CBI is numerically higher than that for SI

20. Post Hoc Outcome: Least Squares Mean Symptom Distress Score on the Outcomes Questionnaire Using a Repeated Measures ANCOVA Adjusted for Baseline Scores and Time Effects
Description: The Symptom Distress subscale assesses symptoms of affective disorders, anxiety disorders, adjustment disorders and stress related illness. It consists of 25 items, with a score range from 0 to 100. Higher scores indicate more symptoms and distress.
Time Frame: Baseline, week 12 (end of treatment), 3 and 6 months post-treatment
Population: Participants were randomly assigned to CBI or SI. Those with one or more post-baseline assessments (wk 12, 3- and/or 6-mo follow-up) were included in HLM analyses. Not all participants had post-baseline data, and some who didn't complete treatment had one or more post-baseline measures. Least Square means and differences adjusted for baseline and time effects from repeated measures ANCOVA are shown. Full Information Maximum Likelihood was used to account for missing data.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Cognitive Behavioral Intervention | Supportive Intervention
Number analyzed (Participants) | 26 | 37
score on a scale | 35.29 (2.56) | 41.58 (2.08)
Statistical Analysis 1: Comparison: Cognitive Behavioral Intervention vs Supportive Intervention; All randomized participants with at least one post-baseline assessment (12 week (end of treatment), 3 mo and/or 6 mo follow-up) were included in the HLM analysis. Full Information Maximum Likelihood was used to account for missing data; Test type: Superiority; p = 0.060, ANCOVA — Threshold for significance was 0.025; Hierarchical Linear Model (HLM) Repeated Measures Analysis of Covariance, controlling for baseline score; Least Squares Mean Difference = -6.29, 95% CI 2-sided [-12.85 to 0.27]; A negative difference means that the adjusted mean for CBI is numerically lower than that for SI, indicating less symptomatic distress

21. Post Hoc Outcome: Least Squares Mean Interpersonal Relations Scale Score on the Outcomes Questionnaire Using a Repeated Measures ANCOVA Adjusted for Baseline Scores and Time Effects
Description: The OQ Interpersonal Relations subscale assesses complaints such as loneliness, conflicts with others, family and marriage problems. High scores reflect more difficulties in these areas. This subscale contains 11 items with a range of 0 to 44.
Time Frame: Baseline, Week 12 (End of Treatment), 3 and 6 months post-treatment
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Cognitive Behavioral Intervention | Supportive Intervention
Number analyzed (Participants) | 26 | 37
score on a scale | 14.66 (1.09) | 17.93 (0.86)
Statistical Analysis 1: Comparison: Cognitive Behavioral Intervention vs Supportive Intervention; [analysis description as in outcome 20, analysis 1]; Test type: Superiority; p = 0.023, ANCOVA — Threshold for significance was 0.025; Hierarchical Linear Model (HLM) Repeated Measures Analysis of Covariance, controlling for baseline score; Least Squares Mean Difference = -3.271, 95% CI 2-sided [-6.083 to -0.458] — A negative difference means that the adjusted mean for CBI is numerically lower than that for SI

22. Post Hoc Outcome: Mean Social Role Scale on the Outcomes Questionnaire Using a Repeated Measures ANCOVA Adjusted for Baseline Scores and Time Effects
Description: The Social Role scale measures the extent to which difficulties in the social roles of worker, homemaker, or student are present. This subscale contains 9 items with a range of 0 to 36. Higher scores indicate more conflicts at work, overwork, distress, and inefficiency in these roles.
Time Frame: Baseline, Week 12 (End of Treatment), 3 and 6 months post-treatment.
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Cognitive Behavioral Intervention | Supportive Intervention
Number analyzed (Participants) | 26 | 37
units on a scale | 11.39 (0.82) | 12.68 (0.67)
Statistical Analysis 1: Comparison: Cognitive Behavioral Intervention vs Supportive Intervention; [analysis description as in outcome 20, analysis 1]; Test type: Superiority; p = 0.23, ANCOVA — Threshold for significance was 0.025; Hierarchical Linear Model (HLM) Repeated Measures Analysis of Covariance, controlling for baseline score; Least Squares Mean Difference = -1.28, 95% CI 2-sided [-3.39 to 0.82] — A negative difference means that the adjusted mean for CBI is numerically lower than that for SI

ADVERSE EVENTS:
Time Frame: 4 years
Arm/Group | Cognitive Behavioral Intervention | Supportive Intervention
All-Cause Mortality (participants affected / at risk) | 1/47 | 1/45
Serious Adverse Events (participants affected / at risk) | 3/47 | 1/45
Other Adverse Events (participants affected / at risk) | 0/47 | 0/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cognitive Behavioral Intervention (N=47) | Supportive Intervention (N=45)
Panic Attack (Psychiatric disorders) | 2 (2) | 0 (0) — Panic Attack
Death (Cardiac disorders) | 1 (1) | 0 (0) — Cardiac attack
Death (Psychiatric disorders) | 0 (0) | 1 (1) — Veteran accidentally overdosed on cocaine and fentanyl

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-11-28): https://cdn.clinicaltrials.gov/large-docs/79/NCT02157779/Prot_SAP_000.pdf
  • Informed Consent Form (2017-09-18): https://cdn.clinicaltrials.gov/large-docs/79/NCT02157779/ICF_001.pdf